CLINICAL TRIAL: NCT04443907
Title: A First-in-patient Phase I/II Clinical Study to Investigate the Safety, Tolerability and Efficacy of Genome-edited Hematopoietic Stem and Progenitor Cells in Subjects With Severe Complications of Sickle Cell Disease
Brief Title: Study of Safety and Efficacy of Genome-edited Hematopoietic Stem and Progenitor Cells in Sickle Cell Disease (SCD)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision of early termination was made due to business reasons and was not a consequence of any safety concern.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CADPT03A12101
Record Dates: First submitted 2020-04-29; First posted 2020-06-23 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
Keywords: Gene therapy; genome-edited hematopoietic stem and progenitor cellular therapy; sickle cell; autologous transplant; BCL11A
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Masking Description: The is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OTQ923 (Experimental): Single intravenous infusion of OTQ923 Part A - Adults treated with OTQ923; Part B - Children age 2-17 treated with OTQ923 based on review of data from Part A by Health agency after a formal interim analysis.
  Interventions: Biological: OTQ923

INTERVENTIONS:
Biological: OTQ923 — Single intravenous infusion of OTQ923 cell suspension
  Other Names: Adult Part A
Biological: OTQ923 — Single intravenous infusion of OTQ923, based on review of data from Part A by Health agencies after a formal interim analysis
  Other Names: Children 2-17 years old - Part B

SUMMARY:
This study evaluated a genome-edited, autologous, hematopoietic stem and progenitor cell (HSPC) product - OTQ923 to reduce the biologic activity of BCL11A, increasing fetal hemoglobin (HbF) and reducing complications of sickle cell disease.

DETAILED DESCRIPTION:
CADPT03A12101 was a multicenter, multi-part, first-in-human, proof-of-concept, open label non-randomized, clinical study in Sickle Cell Disease (SCD) subjects. This study included apheresis of mobilized hematopoietic stem and progenitor cells (HSPCs), ex vivo CRISPR/Cas9-mediated genome editing and expansion, followed by myeloablative conditioning and autologous hematopoietic stem cell transplant (HSCT) with follow-up for a minimum of one year and up to two years.

The study was divided into the following parts:

* Part A - Adult subjects were dosed with OTQ923.
* Part B - Assessment of OTQ923 in pediatric patients, however Part B was not opened.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age 2-40 years inclusive
2. Confirmed diagnosis of sickle cell disease with globin typing (e.g. HbSS, HbSC, HbS/β0-thalassemia or others)
3. Performance status >70% (Karnofsky for subjects >16 years of age and Lansky for subjects <16 years of age)
4. At least one of the following indicators of disease severity as defined in the protocol - Vaso-occlusive pain crisis, Acute chest syndrome, Recurrent priapism, prior stroke, receive chronic transfusions, Red cell alloimmunization
5. Subjects, who have failed, not tolerated or refused hydroxyurea therapy.

Exclusion Criteria:

1. Available matched related donor for HSCT
2. Clinically significant active infection
3. Seropositive for HIV or HTLV
4. Active known malignancy, myelodysplasia, abnormal cytogenetics or immunodeficiency
5. Prior HSCT or gene therapy
6. Known hepatic cirrhosis, bridging hepatic fibrosis or active hepatitis
7. Protocol defined iron overload
8. Cerebrovascular procedure within one year, including pial synangiosis for Moyamoya
9. Severe or progressive arteriopathy or cerebrovascular disease, including Moyamoya

Other protocol defined inclusion/exclusion criteria may apply

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and serious adverse events | up to 24 months
  Number of participants with adverse events (AEs) and serious adverse events (SAEs), including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs.
Fetal hemoglobin (HbF) expression 6 months after hematopoietic stem cell transplant (HSCT) | at 6 months
  Assessment of HbF expression will be done by measuring total fetal hemoglobin over time.
Time to reach absolute neutrophil count (ANC) ≥500/μL for 3 consecutive days | up to 24 months
  Time to engraftment is defined as first of 3 consecutive days when an absolute neutrophil count (ANC) ≥500/μL after receiving OTQ923 was reached.

SECONDARY OUTCOMES:
Durability of hematologic engraftment | up to 24 months
  Engraftment durability/persistence by measuring the proportion of alleles with on-target CRISPR modification in peripheral blood (total white blood cells (WBC)) and bone marrow over time up to 24 months
Proportion of subject to achieve 30% of total HbF at 12 months | 12 months
  Assessment of HbF expression will be done by measuring total fetal hemoglobin over time.
Time to achieve 30% total HbF | up to 24 months
  Assessment of HbF expression will be done by measuring total fetal hemoglobin over time.
Time to peak total HbF | up to 24 months
  Assessment of HbF expression will be done by measuring total fetal hemoglobin over time.
Percentage of edited WBC and bone marrow cells by time points | up to 24 months
  Assessment of in vivo cellular kinetics
Number of participants with treatment induced anti-Cas9 humoral and cellular immunogenicity | up to 24 months
  To evaluate presence of pre-existing or treatment induced anti-Cas9 humoral and cellular immunogenicity
Overall Survival | up to 24 months
  To evaluate the overall survival which is defined as the time from date of start of treatment to date of death to any cause.
Transplant-related mortality | up to 24 months
  Assessment of mortality
Evaluation of effect on patient-reported outcomes from baseline and post-HSCT with age appropriate patient reported measures | up to 24 months
  Determine health status following instruments ASCQ-ME emotional impact
Number of participants with change from baseline of annualized VOC rate by 65% | Baseline, 12 months
  The annualized rate at baseline will be compared to that of vaso-occlusive crises (VOC) at 12 months.
Number of participants with change from baseline of annualized SCD complications (aggregate of VOC, ACS, priapism and stroke) and if relevant, rate of transfusion by 65% | Bseline, 12 months
  The annualized rate at baseline will be compared to that of aggregate Sickle Cell Disease (SCD) complications (VOC, acute chest syndrome (ACS), priapism, and stroke) and transfusions at 12 months.
Evaluation of effect on patient-reported outcomes from baseline and post-HSCT with age appropriate patient reported measures | up to 24 months
  Determine health status following instruments PROMIS fatique
Evaluation of effect on patient-reported outcomes from baseline and post-HSCT with age appropriate patient reported measures | up to 24 months
  Determine health status following instruments PROMIS physical functioning
Evaluation of effect on patient-reported outcomes from baseline and post-HSCT with age appropriate patient reported measures | up to 24 months
  Determine health status following instruments ASCQ-ME sleep impact
Evaluation of effect on patient-reported outcomes from baseline and post-HSCT with age appropriate patient reported measures | up to 24 months
  Determine health status following instruments ASCQ-ME pain impact

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - St Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Ligon JA, Cupit-Link MC, Yu C, Levine J, Foley T, Rotz S, Sharma A, Gomez-Lobo V, Shah NN. Pediatric Cancer Immunotherapy and Potential for Impact on Fertility: A Need for Evidence-Based Guidance. Transplant Cell Ther. 2024 Aug;30(8):737-749. doi: 10.1016/j.jtct.2024.06.006. Epub 2024 Jun 10. PMID 38866240
- [Derived] Sharma A, Boelens JJ, Cancio M, Hankins JS, Bhad P, Azizy M, Lewandowski A, Zhao X, Chitnis S, Peddinti R, Zheng Y, Kapoor N, Ciceri F, Maclachlan T, Yang Y, Liu Y, Yuan J, Naumann U, Yu VWC, Stevenson SC, De Vita S, LaBelle JL. CRISPR-Cas9 Editing of the HBG1 and HBG2 Promoters to Treat Sickle Cell Disease. N Engl J Med. 2023 Aug 31;389(9):820-832. doi: 10.1056/NEJMoa2215643. PMID 37646679
- [Derived] Sharma A, Young A, Carroll Y, Darji H, Li Y, Mandrell BN, Nelson MN, Owens CL, Irvine M, Caples M, Jerkins LP, Unguru Y, Hankins JS, Johnson LM. Gene therapy in sickle cell disease: Attitudes and informational needs of patients and caregivers. Pediatr Blood Cancer. 2023 Jun;70(6):e30319. doi: 10.1002/pbc.30319. Epub 2023 Mar 28. PMID 36975201
- [Derived] Persaud Y, Mandrell BN, Sharma A, Carroll Y, Irvine M, Olufadi Y, Kang G, Hijano DR, Rai P, Hankins JS, Johnson LM. Attitudes toward COVID-19 vaccine among pediatric patients with sickle cell disease and their caregivers. Pediatr Blood Cancer. 2023 May;70(5):e30274. doi: 10.1002/pbc.30274. Epub 2023 Mar 1. PMID 36860093
- [Derived] Bhoopalan SV, Yen JS, Levine RM, Sharma A. Editing human hematopoietic stem cells: advances and challenges. Cytotherapy. 2023 Mar;25(3):261-269. doi: 10.1016/j.jcyt.2022.08.003. Epub 2022 Sep 17. PMID 36123234
- See also: CADPT03A12101 Clinical Trial Results Form — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18388
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=3121